CLINICAL TRIAL: NCT05981092
Title: A PROSPECTIVE MULTINATIONAL STUDY OF THE NATURAL HISTORY OF PARTICIPANTS WITH BAG3 MUTATION ASSOCIATED DILATED CARDIOMYOPATHY
Brief Title: A Study About the Natural History in Adults With BAG3 Dilated Cardiomyopathy (a Type of Heart Disease) (BAG3 DCM)
Status: Active, not recruiting | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: R0765C00001; C4981001 (Other: Alexion); ALXN2350-DCM-501 (Other: Alexion)
Record Dates: First submitted 2023-06-14; First posted 2023-08-08 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Cardiomyopathy, Dilated; Bcl-2 Anathogene-3 (BAG3) Dilated Cardiomyopathy (DCM)
Keywords: BAG3; DCM; cardiomyopathy; dilated cardiomyopathy; heritable heart disease; heart disease
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathies; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAG3 DCM: A single arm observational trial where all participants will undergo the same schedule of assessments.

SUMMARY:
The purpose of this study is to learn about the natural progression of DCM (dilated cardiomyopathy) caused by BAG3 gene mutations. DCM is a condition as the heart muscle is weakened and the heart becomes enlarged. This makes it hard for the heart to pump enough blood for the body.

The study is seeking up to about 35 participants who have:

* BAG3 mutation (change in the gene) that causes or is likely to cause dilated cardiomyopathy
* NYHA (New York Heart Association) Class I-IV at screening (Stage B-D)
* Left Ventricular Ejection Fraction less than or equal to 50% (meaning reduced heart function)

All participants in this study will receive their usual treatment. The investigators will observe the natural progression of people who have BAG3 DCM. This will help the investigators better understand the disease and aid in future research.

Participants will take part in this study for three years. During this time, participants will visit the site at least 8 times (about every 3 months for the first year and annually during year 2 and three). Participants will undergo study procedures and give information about their health. These procedures will include a physical exam, cardiac magnetic resonance imaging, echocardiography, ECG monitoring, activity monitoring, cardiopulmonary exercise testing, and blood tests. Participants will answer questions about health and quality of life. The study team will also call participants about 1 time over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Documented BAG3 mutation that causes or is likely to cause dilated cardiomyopathy
* Heart failure Stage B-D, New York Heart Association (NYHA) Class I-IV
* Left Ventricular Ejection Fraction ≤50% (i.e., Reduced Heart Function)

Exclusion Criteria:

* Acute decompensated heart failure within 1 month prior to enrollment.(such as hospitalization)
* Any of the following within 3 months prior to screening: myocardial infarction (MI), cardiac surgical procedures (other than for pacemaker/ICD/CRT-defibrillator [CRT-D] implantation), acute coronary syndrome, or hospitalization for cardiac arrhythmia.
* History of heart transplantation
* eGFR <30 mL/min/1.73 m2 (significantly impaired kidney function)
* Noncardiac condition that limits lifespan to <1 year.
* Presence of other form(s) of cardiomyopathy contributing to heart failure
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement).
* No more than 3 first-degree members of the same family who are already participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic and referrals from primary care clinic to investigational sites
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2027-08-12 (Estimated); Study Completion 2027-08-12 (Estimated)

PRIMARY OUTCOMES:
Determine baseline of cardiac structure and function in BAG3 associated DCM. | Baseline
  Baseline measures of left ventricular volumes at end systole and diastole using imaging at baseline.
Determine changes over time in cardiac structure and function in BAG3 associated DCM. | 3 years
  Changes over time of left ventricular volumes at end systole and diastole using imaging over the course of 3 years follow up time.

SECONDARY OUTCOMES:
Change from Baseline in high sensitivity troponin I (hsTNI) levels | Baseline to year 3
  HsTNI will be collected at baseline through 3 years to observe the natural history (baseline and variance) of the biomarker and the correlation of hsTNI to severity of clinical disease progression.
Change from Baseline in high sensitivity troponin T (hsTNT) levels | Baseline to year 3
  HsTNT will be collected at baseline through 3 years to observe the natural history (baseline and variance) of the biomarker and the correlation of hsTNT to severity of clinical disease progression.
Change from Baseline in N-terminal Prohormone of Pro-Brain-Type Natriuretic peptide (NT-proBNP) levels | Baseline to year 3
  NT-proBNP will be collected at baseline through 3 years to observe the natural history (baseline and variance) of the biomarker and the correlation of NT-proBNP to severity of clinical disease progression.
Change from baseline in Measures of Oxygen Capacity | Baseline to year 3
  Measured via Cardio Pulmonary Exercise Testing (CPET).
Change from Baseline in Scores of Kansas City Cardiomyopathy Questionnaire (KCCQ) domains | Baseline to year 3
Change from Baseline in Scores of Patient Global Impression of Severity (PGI-S) | Baseline to year 3
Change from Baseline in Scores of Patient Global Impression of Change (PGI-C) | Baseline to year 3
Define the rate of cardiac status changes over time. | 3 years
  The frequency and rate of incidence of death, heart transplant, MCS, heart failure, hospitalization, appropriate implantable cardioverter defibrillator shock, or aborted SCD.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (6):
  - Research Site, Palo Alto, California
  - Research Site, Aurora, Colorado
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, The Bronx, New York
  - Research Site, Philadelphia, Pennsylvania
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Maastricht
- Research Site, Warsaw, Poland
- Spain (4):
  - Research Site, Majadahonda, Madrid
  - Research Site, El Palmar, Murcia
  - Research Site, A Coruña
  - Research Site, Madrid
- United Kingdom (2):
  - Research Site, Harefield, London
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR